CLINICAL TRIAL: NCT05354414
Title: A Randomized Crossover Pragmatic Study to Evaluate Virtual Reality for the Mitigation of Anxiety During Intrathecal Administration in Patients With Spinal Muscular Atrophy. REALITY Study.
Brief Title: Virtual Reality for the Mitigation of Anxiety During Intrathecal Administration in Participants With Spinal Muscular Atrophy
Acronym: REALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FR-NMD-12094
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR followed by SOC (Experimental): Participants will receive a 20-minute (min) VR session at the first nusinersen IT (IT1), followed by SOC (local anesthesia - lidocaine or intravenous sedation) at the subsequent nusinersen IT (IT2) during the main study, later followed by 20-min VR sessions at two subsequent nusinersen ITs (IT3 and IT4) during the extension period, for up to 450 days.
  Interventions: Device: Virtual reality; Procedure: Standard of Care
- SOC followed by VR (Experimental): Participants will receive SOC (local anesthesia - lidocaine or intravenous sedation) at nusinersen IT1, followed by a 20-min VR session at the subsequent nusinersen IT (IT2) during the main study, later followed by 20-min VR sessions at two subsequent nusinersen ITs (IT3 and IT4) during the extension period, for up to 450 days.
  Interventions: Device: Virtual reality; Procedure: Standard of Care

INTERVENTIONS:
Device: Virtual reality — Administered as specified in the treatment arm.
Procedure: Standard of Care — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of the study is to evaluate anxiety level during intrathecal administration (IT) under standard of care (SOC) and virtual reality (VR) conditions using a reliable self-rating scale.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants aged 7 years and greater
* Genetically documented spinal muscular atrophy linked to chromosome 5q (5q-SMA)
* Loading nusinersen dose period is completed, and ongoing treatment with nusinersen
* Ability of the candidate and/or their legally authorized representatives (e.g., parent, spouse, or legal guardian), as appropriate and applicable, to understand the purpose and risks of the study, to provide informed consent, and to authorize the use of confidential health information in accordance with national and local privacy regulations
* Signed written informed consent from adult participants, or from legal authorized representatives for minors

Key Exclusion Criteria:

* History of any clinically significant abnormalities that would render the candidate unsuitable for VR (e.g., visual or hearing impairment, presence of eye, face or sclap injuries) or for inclusion (e.g. cognitive impairment), as determined by the Investigator
* Conditions that could be exacerbated by the VR environment, such as: (i) current symptomatic nausea, vomiting, dizziness, migraine; (ii) history of psychosis, hallucinations, epilepsy
* Ongoing medical conditions or treatments that according to the Investigator would interfere with the conduct and assessments of the study (e.g. general anesthesia)
* Participants wearing a pacemaker and pregnant woman

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Anxiety (VAS-A) Score During IT as Evaluated by the Participant Just After IT | Up to 450 days
  The VAS-A scale is used in the assessment of anxiety. The 101-point scale (0 to 100) is a horizontal 100 millimeter (mm) line that starts with no anxiety on the left and ends with maximum anxiety on the right. The VAS score is determined by measuring in mm from the left-hand end of the line to the point that the participant marks. High scores on the scale indicate that anxiety is high.

SECONDARY OUTCOMES:
Blood Pressure Before and After IT | Up to 450 days
  Systolic and diastolic blood pressures will be assessed.
Heart Rate Before and After IT | Up to 450 days
Short State-Trait Anxiety Inventory (Short STAI) Score During IT as Evaluated by the Participant Just After IT | Up to 450 days
  The 6-item short form of the Spielberger STAI is used to measure self-reported symptoms of state anxiety. It consists of 6 questions each having scale 1 (Almost Never) to 4 (Almost Always). The score range for the short STAI is 6 to 24 points, with 6 points signifying no anxiety and 24 points signifying the highest level of anxiety.
Number of Participants With Use of Medication/Intervention for Anxiety and Pain Management Before, During and up to 72 hour (h) After IT | Up to 450 days
Visual Analog Scale for Pain (VAS-P) Score Just After IT | Up to 450 days
  The VAS-P scale is used in the assessment of pain. The 101 point scale (0 to 100) is a horizontal 100 mm line that starts with no pain on the left and ends with maximum pain on the right. The VAS score is determined by measuring in mm from the left hand end of the line to the point that the participant marks. High scores indicate worse pain.
Maximal VAS-P Score Within 72h of IT | Up to 450 days
  The VAS-P scale is used in the assessment of pain. The 101 point scale (0 to 100) is a horizontal 100 mm line that starts with no pain on the left and ends with maximum pain on the right. The VAS score is determined by measuring in mm from the left hand end of the line to the point that the participant marks. High scores indicate worse pain.
Number of Participants With Satisfactory Experience of Using VR, Desire to Continue IT, Desire to Continue VR | Up to 150 days
  Participants will be asked to complete a satisfaction survey to evaluate his/her experience. It is a questionnaire consisting of 6 (for age >12 years) to 7 (for age <12 years) questions.
Number of Participants With Satisfactory Experience of Using VR, as Assessed by Custom Care Team | Up to 150 days
  The custom care team will be asked to complete a satisfaction survey to evaluate participant's experience. It is a questionnaire consisting of 5 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- France (12):
  - Chu d' Angers, Angers
  - CHRU de Brest, Brest
  - Chu de Clermont Ferrand, Clermont-Ferrand
  - APHP- Raymond Poincaré Paris, Garches
  - Chu de Lille, Lille
  - CHU Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - Chu de Nice, Nice
  - APHP- Necker Paris, Paris
  - APHP- Trousseau Paris, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/